CLINICAL TRIAL: NCT02395549
Title: A Study to Determine the Efficacy of Topically Applied MTC896 Gel in Subjects With Acne Vulgaris
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mimetica Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCL15001
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 0.375% (w/w) MTC896 Gel (Experimental): 0.375% (w/w) MTC896 Gel will be applied bid to the whole face for 12 weeks.
  Interventions: Drug: 0.375% (w/w) MTC896 Gel
- 0.75% (w/w) MTC896 Gel (Experimental): 0.75% (w/w) MTC896 Gel will be applied bid to the whole face for 12 weeks.
  Interventions: Drug: 0.75% (w/w) MTC896 Gel
- 1.5% (w/w) MTC896 Gel (Experimental): 1.5% (w/w) MTC896 Gel will be applied bid to the whole face for 12 weeks.
  Interventions: Drug: 1.5% (w/w) MTC896 Gel
- Vehicle Control Gel (Placebo Comparator): Vehicle Control Gel will be applied bid to the whole face for 12 weeks.
  Interventions: Drug: Vehicle Control Gel

INTERVENTIONS:
Drug: 0.375% (w/w) MTC896 Gel — 0.375% (w/w) MTC896 Gel
  Arms: 0.375% (w/w) MTC896 Gel
Drug: 0.75% (w/w) MTC896 Gel — 0.75% (w/w) MTC896 Gel
  Arms: 0.75% (w/w) MTC896 Gel
Drug: 1.5% (w/w) MTC896 Gel — 1.5% (w/w) MTC896 Gel
  Arms: 1.5% (w/w) MTC896 Gel
Drug: Vehicle Control Gel
  Arms: Vehicle Control Gel

SUMMARY:
This study is designed to investigate the efficacy, safety and tolerability of MTC896 Gel in subjects with acne. In this study, MTC896 Gel will be applied at 3 concentrations, twice daily (bid) for 12 weeks and compared against a vehicle control.

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or nonpregnant, non-lactating, non-breastfeeding female, 16 to 65 years of age, inclusive, at the time of screening;
2. Has provided written informed consent/assent (which includes consent for photographs, if applicable, to be taken at Baseline and end-of-treatment/end-of-study [EOT/EOS] visits);
3. Has been diagnosed with mild-to-severe acne vulgaris defined as:

   * At least 20 inflammatory lesions,
   * At least 20 noninflammatory lesions,
   * ≤ 2 nodular lesions, and
   * Investigator Global Assessment of 2 or greater;
4. Is willing to comply with the requirements of the protocol;
5. If female and of child-bearing potential or premenarcheal, has a negative urine pregnancy test at Screening and Baseline / Day 1 and is willing to use effective contraception during the study and for 30 days after the last study medication application. Females are considered to be of childbearing potential unless surgically sterilized (hysterectomy, bilateral oophorectomy, tubal ligation), diagnosed as infertile, or are postmenopausal for at least 1 year; (Acceptable methods of birth control are defined as: abstinence, oral contraceptives, contraceptive patches/implants, Depo-Provera®, double barrier methods (e.g. condom and spermicide) or an intrauterine device (IUD). Birth control method must have been stable/unchanged for 12 weeks prior to Baseline and must remain unchanged during study participation);
6. If male, has been vasectomized or agrees to use an accepted method of birth control with female partner during study participation and for 30 days after the last study medication application;
7. Is in good health and free from any disease which, in the opinion of the Investigator, would put the subject at risk if participating in the study;
8. Is free of any systemic or dermatologic disorder, which, in the opinion of the Investigator, will interfere with the study results or increase the risk of adverse events;
9. Is willing to abstain from using any facial treatment products on the face during the study (continued use of make-up is permitted but may not be changed within 2 weeks prior to the study period or during the entire study period);
10. Is willing to avoid sun exposure and to protect the face with a hat/visor; sunscreen use is recommended/allowed when sun exposure cannot be avoided;
11. If male, must agree to shave the treatment area and must agree not to alter his routine shaving regimen for the duration of the study;
12. Is willing to refrain from using any treatments, other than the study medication, including antibiotics, for acne present on the face. Topical acne treatments that do not have significant or measurable systemic absorption (e.g. benzoyl peroxide, salicylic acid) are allowed for treatment of acne of the back, shoulders, and chest only.

Exclusion Criteria:

1. People who would otherwise qualify for the study, but are living in the same household as a study subject, are not allowed to participate in the study;
2. Pregnant or lactating or plan to become pregnant within 1 month (30 days) of study completion;
3. Known allergy/sensitivity to any of the study medication components;
4. Any skin condition which may interfere with the evaluation of safety or of acne vulgaris (e.g. rosacea, seborrheic dermatitis, perioral dermatitis, corticosteroid-induced acne or folliculitis);
5. Excessive facial hair that would interfere with diagnosis or assessment of acne vulgaris;
6. Excessive sun exposure, in the opinion of the Investigator, or use of tanning booths;
7. Active cystic acne or acne conglobata, acne fulminans, and secondary acne;
8. Screening clinical chemistry or hematology laboratory value that is considered clinically significant, in the opinion of the Investigator;
9. Participation in an investigational drug study within 30 days prior to Screening;
10. Is a poor medical risk because of other systemic diseases or active uncontrolled infections, in the opinion of the Investigator;
11. Any other condition which, in the judgment of the Investigator, would put the subject at unacceptable risk for participation in the study;
12. Within 9 months (270 days) prior to Baseline and throughout the study:

    - Oral retinoid use (e.g. isotretinoin);
13. Within 6 months (180 days) prior to Baseline and throughout the study:

    - Treatment with Vitamin A supplements greater than 10,000 units/day;
14. Within 3 months (90 days) prior to Baseline and throughout the study:

    * Use of androgen receptor blockers (such as spironolactone or flutamide);
    * Initiation of treatment with hormonal therapy or dose change to hormonal therapy;
    * Dose and frequency of use of any hormonal therapy started more than 3 months (90 days) prior to Baseline must remain unchanged throughout the study;
    * Hormonal therapies include, but are not limited to, testosterone, anabolic steroids, birth control pills;
15. Within 8 weeks (56 days) prior to Baseline and throughout the study:

    - Facial procedures (chemical or laser peel, microdermabrasion, etc.);
16. Within 4 weeks (28 days) prior to Baseline and throughout the study:

    * Treatment with systemic corticosteroids (including intranasal and inhaled corticosteroids);
    * Treatment with systemic antibiotics or systemic anti-acne drugs or systemic anti-inflammatory drugs; Note: Non-steroidal anti-inflammatory drugs (NSAIDs) and aspirin use on an as-needed basis and if not used consecutively for >14 days prior to Baseline is acceptable and does not require washout. Low dose (81 mg) aspirin taken daily is acceptable.
    * Prescription topical retinoid use on the face (e.g. tretinoin, tazarotene, adapalene);
    * Antifungals, antiretrovirals and antibiotics included in the CYP 3A4 and CYP 3A5;
17. Within 2 weeks (14 days) prior to Baseline and throughout the study:

    * Treatment with topical prescription antibiotics (e.g. dapsone, clindamycin, erythromycin, or sulfacetamide);
    * Treatment with over-the-counter (OTC) topical medications for the treatment of acne vulgaris including benzoyl peroxide, topical anti-inflammatory medications, corticosteroids, α-hydroxy/glycolic acid on the face;
18. Within 1 day prior to Baseline and throughout the study:

    * Grapefruit juice which is included in the CYP 3A4 and CYP 3A5.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Absolute change from baseline in inflammatory lesion counts | Week 12
Absolute change from baseline in noninflammatory lesion counts | Week 12
Proportion of subjects with Investigator"s Global Assessment (IGA) success | Week 12
  i.e., who achieved a minimum 2-grade improvement from baseline

SECONDARY OUTCOMES:
Percent change from baseline in inflammatory lesion counts | Weeks 4, 8 and 12
Percent change from baseline in noninflammatory lesion counts | Weeks 4, 8 and 12
Percent change from baseline in total lesion counts | Weeks 4, 8 and 12
Absolute change from baseline in inflammatory lesion counts | Weeks 4 and 8
Absolute change from baseline in noninflammatory lesion counts | Weeks 4 and 8
Absolute change from baseline in total lesion counts | Weeks 4, 8 and 12
Proportion of subjects with IGA success | Weeks 4 and 8
  i.e. who achieved a minimum 2-grade improvement from baseline
Time to IGA success | Week 12
Proportion of subjects who achieved at least a 2 grade reduction and an IGA score of clear or almost clear | Weeks 4, 8 and 12
Proportion of subjects who achieved a "Clear" or "Almost Clear" IGA score | Weeks 4, 8 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Debra Dow, Study Director — Symbio, LLC
Locations (19):
- United States (19):
  - Sacramento, California
  - San Diego, California
  - Denver, Colorado
  - Sanford, Florida
  - West Palm Beach, Florida
  - Louisville, Kentucky
  - Warren, Michigan
  - Minneapolis, Minnesota
  - Albuquerque, New Mexico
  - High Point, North Carolina
  - Hershey, Pennsylvania
  - Johnston, Rhode Island
  - Warwick, Rhode Island
  - Nashville, Tennessee
  - Austin, Texas
  - College Station, Texas
  - Plano, Texas
  - Salt Lake City, Utah
  - Spokane, Washington